CLINICAL TRIAL: NCT04761705
Title: A Phase 1/2 Safety and Efficacy Study of JV-GL1 Applied to the Periorbital Skin in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Safety and Efficacy Study of JV-GL1 in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Awaiting transition to Part 2
Sponsor: JeniVision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JV-GL1-OCU-GL-101/201-01
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Ocular Hypertension; Open Angle Glaucoma
Keywords: open angle glaucoma; Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle | interventions — Latanoprost; Ophthalmic Solutions

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Randomized Part 2, Arm 1 (Experimental): Dose 1 selected in Part I
  Interventions: Drug: JV-GL1
- Randomized Part 2, Arm 2 (Experimental): Dose 2 selected in Part I
  Interventions: Drug: JV-GL1
- Randomized Part 2, Arm 3 (Active Comparator)
  Interventions: Drug: Latanoprost 0.005% Ophthalmic Solution

INTERVENTIONS:
Drug: JV-GL1 — Experimental Treatment
  Arms: Randomized Part 2, Arm 1; Randomized Part 2, Arm 2
Drug: Latanoprost 0.005% Ophthalmic Solution — Active Control
  Arms: Randomized Part 2, Arm 3

SUMMARY:
The aim of this research study is to assess the safety and feasibility of lowering intraocular pressure (IOP) using an experimental study drug, JV-GL1.

DETAILED DESCRIPTION:
This is an open-label, dose escalation and dose expansion, study in adult participants with open-angle glaucoma or ocular hypertension. The study is divided into 2 parts:

Part 1 of the study is a dose escalation, sequentially testing escalating doses of JV-GL1.

Part 2 of the study will be randomized 2:2:1 (Experimental Dose A: Experimental Dose B: Active Control), treating additional subjects at the selected JV-GL1 doses or Latanoprost for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* bilateral open-angle glaucoma or ocular hypertension

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure (IOP) | From Baseline to Day 28 of Treatment
  Change from baseline in Intraocular Pressure (IOP)

CONTACTS AND LOCATIONS:
Overall Officials: David Wirta, MD, Principal Investigator — Eye Research Foundation, Inc.
Locations (1):
- Eye Research Foundation, Newport Beach, California, United States